CLINICAL TRIAL: NCT02683876
Title: Metabolomic Profiling of Urine Samples for the Identification of Novel Biomarkers and Mechanisms in the Diagnosis and Management of Malodor Associated With Metabolic Inefficiencies
Brief Title: Exploratory Study of Relationships Between Malodor and Urine Metabolomics
Status: Completed | Type: Observational
Sponsor: Mebo Research, Inc. (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: 201505010014MEBO
Record Dates: First submitted 2016-02-03; First posted 2016-02-17 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: body odor, malodor, halitosis
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Body Odor; Halitosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subjects with malodor: individuals with self-reported odor issues suspected to be associated with microbial imbalance on or inside the body and inefficient metabolism as evidenced from other laboratory tests
- Healthy control: individuals not complaining of uncontrollable or unpredictable malodor episodes

SUMMARY:
The purpose of this study is to identify metabolic signatures associated with malodor conditions. The investigators will perform state-of-the art metabolomics tests and bioinformatic data mining to explore if conditions leading to malodor can be screened by metabolomic profiling of urine samples.

DETAILED DESCRIPTION:
In this study, metabolite profiling analysis will be carried out on urine samples of individuals with malodor conditions related to metabolism inefficiencies. Metabolic profiles will be identified using the metabolomics equipment located in the NMR, HPLC and MS facilities of the Metabolomics Innovation Centre (TMIC). Multivariate statistical analyses will be used, as well as other approaches to mine complex data from heterogeneous sources.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* unpredictable and uncontrollable episodes of malodor
* willing and able to ship a urine sample (in the kit provided) by an overnight courier to Edmonton, Alberta, Canada
* good general health

Exclusion Criteria:

* serious medical conditions that require treatment
* conditions that, in the opinion of the investigator, would prevent participation
* under the age of 18
* elect not to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals complaining of uncontrollable episodes of malodor suspected to be caused by inefficient body metabolism
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wishart, PhD, Principal Investigator — The Metabolomics Innovation Centre (TMIC); Irene Gabashvili, PhD, Principal Investigator — MeBo Research
Locations (2):
- MeBO Research, Miami, Florida, United States
- The Metabolomics Innovation Centre, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
to prevent risks of re-identification.

REFERENCES:
- [Background] Emwas AH, Roy R, McKay RT, Ryan D, Brennan L, Tenori L, Luchinat C, Gao X, Zeri AC, Gowda GA, Raftery D, Steinbeck C, Salek RM, Wishart DS. Recommendations and Standardization of Biomarker Quantification Using NMR-Based Metabolomics with Particular Focus on Urinary Analysis. J Proteome Res. 2016 Feb 5;15(2):360-73. doi: 10.1021/acs.jproteome.5b00885. Epub 2016 Jan 20. PMID 26745651
- [Result] I.S. Gabashvili. Identifying subtypes of a stigmatized medical condition medRxiv 19005223; doi: https://doi.org/10.1101/19005223
- See also: The Metabolomics Innovation Centre (TMIC) — https://www.metabolomicscentre.ca/
- See also: MeBO Research — https://meboresearch.org/
- See also: Gabashvili, I.S. NCT02683876: Documentation of Clinical Trial Data and Procedures. — https://aurametrix.com/NCT2683876

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Malodor: individuals with self-reported socially debilitating odor episodes
Period: Overall Study
Arm/Group | Subjects With Malodor | Healthy Control
Started | 17 | 22
Completed | 15 | 22
Not Completed | 2 | 0
Not completed — samples damaged during shipping | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With Malodor | Healthy Control | Total
Number analyzed (Participants) | 17 | 22 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 21 | 38
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 5 | 14 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 17 | 22 | 39
Metabolites measured in urine samples [Count of Participants; unit: Participants] | 15 | 22 | 37

OUTCOME MEASURES:

1. Primary Outcome: Differences in Metabolite Concentrations in Urine Between Individuals With Malodor Issues and Age-matched Healthy Controls.
Description: The investigators would like to validate if urine metabolomic profiling can be used for identifying key metabolomic signatures associated with malodor.
  Differences in metabolite concentrations will be measured by mass spectrometry, to compare urine samples from individuals with malodor issues, and age-matched healthy controls.
Time Frame: time from diagnostic urine sample collection to dispatch of results
Measure: Mean (Full Range); unit: uMol/mM creatinine
Arm/Group | Subjects With Malodor | Healthy Control
Number analyzed (Participants) | 15 | 22
uMol/mM creatinine
  Arginine | 3.4 [1.3 to 7.9] | 8.6 [1.5 to 18.6]
  Citruline | 0.443 [0.175 to 1.185] | 0.8 [0.2 to 1.7]
  Asymmetric dimethylarginine | 4.0 [2.8 to 7.0] | 3.0 [0.2 to 7.0]
  Dopamine | 0.18 [0.10 to 0.28] | 0.10 [0.066 to 0.30]
  Glycine | 142.5 [45.4 to 283.0] | 101.0 [37.0 to 300.0]
  Histamine | 0.05 [0.016 to 0.15] | 0.03 [0.01 to 0.10]
  3-Hydroxytetradecenoylcarnitine | 0.0080 [0.001 to 0.087] | 0.0020 [0.0008 to 0.0040]
  Lysine | 4.7 [2.3 to 10.3] | 17.9 [3.6 to 56.1]

2. Secondary Outcome: Correlations Between Urine Biomarkers and Frequency/Severity of Malodor Symptoms (Questionnaires)
Description: The investigators will comprehensively analyze the ability of metabolite levels to discriminate frequent and severe from less severe malodor symptoms. The severity of the disease was assessed trough interviews (frequency of key symptoms) and prior laboratory tests.
Time Frame: time from sample collection to notification of results and follow-up needed.
Measure: Mean (Standard Deviation); unit: µmol/mmol creatinine
Groups:
- Subjects With More Severe Disease: More severe form of MEBO based on self-reports and prior tests
- Subjects With Less Severe Disease: Subjects with less severe symptoms based on self-reports
Arm/Group | Subjects With More Severe Disease | Subjects With Less Severe Disease
Number analyzed (Participants) | 9 | 6
µmol/mmol creatinine
  Arginine | 3 (2) | 3 (2)
  Citruline | 0.5 (0.3) | 0.4 (0.3)
  Asymmetric dimethylarginine | 4 (2) | 3 (1)
  Dopamine | 0.2 (0.1) | 0.2 (0.1)
  Glycine | 146 (91) | 121 (90)
  Histamine | 0.06 (0.04) | 0.04 (0.03)
  3-Hydroxytetradecenoylcarnitine | 0.012 (0.028) | 0.002 (0.001)
  Lysine | 5 (3) | 4 (3)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 6 months after sample collection, 1 year after initial enrollment.
Arm/Group | Subjects With Malodor | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/22
Other Adverse Events (participants affected / at risk) | 0/17 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT02683876/Prot_SAP_000.pdf